CLINICAL TRIAL: NCT03289169
Title: A Single-Arm Trial, Open-label, Repeated, Long-term, Multi-center, A Phase IV Clinical Trial to Evaluate the Long-term Efficacy and Safety of Repeat Treatment With MEDITOXIN® in Treatment of Glabella Line
Brief Title: Long-term Safety and Efficacy of MEDITOXIN® in Treatment Glabellar Lines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT01-KR16GBL401
Record Dates: First submitted 2017-09-19; First posted 2017-09-20 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MEDITOXIN (Experimental): Meditoxin(Botulinum toxin type A)
  Interventions: Drug: MEDITOXIN®

INTERVENTIONS:
Drug: MEDITOXIN® — 20U of Meditoxin® is injected to two places on the corrugators muscle for each eye and one place on the procerus muscle, total of 5 sites.
  Other Names: Neuronox®

SUMMARY:
This study evaluates the long-term safety of repeated administrations of Meditoxin® in the treatment of moderate to severe glabellar lines.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 20 and 65
* Patients attaining ≥grade 2 (moderate) in the investigator's rating of the severity of glabella lines at maximum frown
* Patients who can comply with the study procedures and visit schedule
* Patients who voluntarily sign the informed consent

Exclusion Criteria:

* Patients with medical conditions who may be at greater risk due to the administration of the investigational drugs (e.g.. diseases that may affect the neuromuscular action including Myasthenia Gravis, Lambert-Eaton Syndrome, Amyotrophic Lateral Sclerosis and motor neuropathy)
* Patients with the history of facial nerve paralysis or the symptoms of eyelid ptosis
* Patients who have received other procedures which may affect glabellar and forehead lines within 6 months
* Patients who have received other procedures which may affect glabellar and forehead lines within 6 months
* Patients who were injected with botulinum toxin within the past 3 months
* Patients with allergy or hypersensitivity to the investigational drugs or their components
* Patients who have bleeding tendency or taking anti-coagulant
* Female subjects who are pregnant or lactating. Female subjects of childbearing age who have a plan to get pregnant during the study period, or do not use available contraceptive methods (Women of childbearing age should have negative urine pregnancy test results at baseline visit (0 week) prior to the first injection.)
* Patients with skin disorders or infection at the injection site
* Patients who are participating in other clinical trials or have participated in other clinical trials 30 days before screening
* Patients who are unable to communicate or follow the instructions
* Patients who are not eligible for this study based on the judgment of an investigator

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-12-30 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
Glabellar line improvement rate at maximum frown confirmed with investigator's live assessment | 4 weeks after final injection
  improvement are defined as subjects with glabellar line severity of none (0) or mild (1).

SECONDARY OUTCOMES:
Glabellar line improvement rate at maximum frown and rest confirmed with investigator's live assessment | 4 weeks after each injection
  Glabellar line improvement rate at maximum frown and rest confirmed with investigator's live assessment at 4 weeks after each injection
Glabellar line improvement rate at maximum frown and rest confirmed with investigator's photo assessment | 4 weeks after each injection
  Glabellar line improvement rate at maximum frown and rest confirmed with investigator's photo assessment at 4 weeks after each injection

CONTACTS AND LOCATIONS:
Locations (1):
- St. Paul Hospital, Seoul, South Korea